CLINICAL TRIAL: NCT04791124
Title: Assessment of Neural Oscillations in Adult Subjects With Down Syndrome and Typically Developing Subjects in Resting State and While Conducting Cognitive Tasks
Acronym: EEGDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Collaborators: Aelis Farma (Industry); Starlab (Unknown)
Responsible Party: Sponsor
Other Study IDs: IMIMFTCL_EEGDS
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; Electroencephalography; Neural oscillations; Endocannabinoids; Gamma Intertrial Coherence
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Typical Developing Subjects: EEG evaluation of typical developing subjects
  Interventions: Other: Electroencephalography
- Down Syndrome Subjects: EEG evaluation of DS subjects
  Interventions: Other: Electroencephalography

INTERVENTIONS:
Other: Electroencephalography — EEG evaluation Composed by three consecutive tests
  1. Resting state EEG, with either eyes open or closed
  2. Auditory steady-state response (ASSR)
  3. Auditory evoked potential

SUMMARY:
Background:

It has been proposed that a hyperactivity of the endocannabinoids system could be involved in the cognitive deficits involved in Down Syndrome (DS). Hyperactivation of the type-1 cannabinoid (CB1) receptor by exogenous cannabinoids, such as the active principle of cannabis tetrahydrocannabinol (THC), induces several modifications of the electroencephalogram (EEG).

The goal of this study is to compare those CB1-dependent EEG parameters in subjects with DS and age-matched typically developing subjects (TD, control group). These investigations can increase our knowledge of the involvement of the CB1 receptor in DS cognitive deficits and potentially identify biomarkers of target engagement of new therapies of this condition.

Hypothesis:

It was recently showed in pre-clinical DS models that the endocannabinoid system is hyperactivated in the brain and that human adult subjects with DS showed higher plasma concentrations of the main endocannabinoids 2-arachidonoylglycerol (2-AG) and anandamide (N-arachidonoylethanolamine, 2-AEA) as compared with those found in typically developing subjects. Alterations of neural oscillations induced by the consumption of THC preparations are well established and it is hypothesized that they would be similar to those found in subjects with DS.

Objectives:

To assess different neural markers using electroencephalography (EEG) in typically developing subjects and in subjects with DS in resting state and while conducting selected cognitive tasks.

Methods:

Non-interventional, cross-sectional, monocenter study in male and female adult subjects with DS and typically developing subjects (total n=48).

ELIGIBILITY:
Common Inclusion Criteria:

* Weight ≥ 50 kg and ≤ 100 kg
* Body mass index (BMI) ≥ 18.5 and ≤ 30

TD group additional Inclusion Criteria:

* Abstinence for alcohol 72h prior to the screening
* Able to read Spanish and adhere to study requirements.
* Signed informed consent prior to any study-mandated procedure.

DS group additional Inclusion Criteria:

* Clinical diagnosis of Down syndrome (full trisomy 21 and translocations) documented by chromosomal analysis (karyotyping).
* Subject understands and accepts the trial procedures.
* Subject assenting and/or willing to participate.
* Signed informed consent by subject and legal representative prior to any study-mandated procedure.
* Subject independently mobile and have sufficient vision and hearing to participate in study evaluations.
* Abstinence for alcohol 72h prior to the screening.
* Clinical Evaluation of Language Fundamentals Preschool-2 (CELF Preschool-2) test score ≥ 7.
* Subjects must have a parent, or other reliable caregiver who agrees to accompany the subject to all clinic visits, provide information about the subject as required by the protocol, and ensure compliance with study tests.
* Subjects are expected to complete all procedures scheduled during the study visits. They must be able to be understood most of the time and must not use other forms of communication, signs, symbol boards or devices as their primary form of communication.

TD group Exclusion Criteria:

* Substance use disorders except for mild alcohol use disorder and/or mild or moderate nicotine use disorder.
* Testing positive for drugs of abuse in urine at screening or the observation day.
* Lifetime clinically significant cardiovascular, renal, pulmonary, hepatic, onco-hematological, endocrine, gastrointestinal, mental or neurological disease.
* Any other diseases or conditions that in the judgment of the investigator would interfere with the subject's ability to comply with study procedures or requirements and/or study results interpretation.
* Any clinically significant findings in physical examination including vital signs.
* Any prescription or over the counter drug (except occasional use of paracetamol) in the last 2 weeks before Day 1 of each period.
* Patient included in a clinical study with drugs in the last three months.

DS group Exclusion Criteria:

* Mosaic Down syndrome
* Personal history of infantile spasms/convulsions/epilepsy, severe head trauma or central nervous system infections (e.g. meningitis), with the exception of a single isolated febrile seizure.
* Subjects with a current Diagnostic of autism spectrum disorder or any primary psychiatric diagnosis. Diagnoses that are secondary, such as attention deficit hyperactivity disorder, depressive disorders and conduct disorders are allowed as long as they are considered to not interfere with study conduct and are stable during the 3 months preceding randomization. Related allowed treatments must be on stable dosing for the last 3 months.
* Symptoms of early dementia as assessed by the Dementia Screening Questionnaire for Individuals with Intellectual Disabilities.
* Substance use disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria.
* Positive urine test for drugs of abuse or alcohol breath test at screening and prior to dosing.
* Epileptiform abnormalities (excluding isolated sharp waves and beyond those expected for age) in 10 min EEG.
* Any life-threatening disease.
* Any other clinically relevant concomitant disease or condition or finding at screening that in the judgment of the investigator could interfere with, the treatment thereof might interfere with, the conduct of the study and related procedures and/or might bias the study results interpretation, or could jeopardize the subject's safety.
* Neuroleptic drugs within 3 months prior to randomization.
* Any clinically significant findings in physical examination including vital signs.
* Any new prescription or over the counter drug (except occasional use of paracetamol) in the last 2 weeks before Day 1 of each period.
* Testing positive for drugs of abuse in urine at screening or the observation day
* Patient included in a clinical study with drugs in the last three months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 24 healthy subjects (12 male and 12 female) with a range age ≥ 18 and ≤ 35 years will be recruited from the typical developing population. A total of 24 healthy subjects (12 male and 12 female) with Down syndrome with a range age ≥ 18 and ≤ 35 years will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Differences in gamma intertrial coherence and power between DS and TD group | During EEG
  Variations in gamma intertrial coherence (ITC) and power during an auditory steady-state response (ASSR) at 40Hz in DS compared to TD subjects.
Differences in power of neural oscillations between DS and TD group | During resting state eyes-closed EEG
  Variations in power of neural oscillations in resting state eyes-closed EEG (alpha, delta, theta, beta, gamma) in DS compared to TD subjects.
Differences in amplitude and latency of various EEG waves between DS and TD group | During EEG while performing a three-stimulus auditory oddball task
  Variations in amplitude and latency of the P300a and P300b, P300, N100 and N200 waves assessed by a three-stimulus auditory oddball task in DS compared to TD subjects.
Differences in EEG complexity between DS and TD group | During EEG
  Variations in EEG complexity measured by the Lempel-Ziv complexity in DS compared to TD subjects.
Differences in EEG brain connectivity, interhemispheric and frontoparietal connectivity, characteristic path and clustering coefficient between DS and TD group | During resting state eyes-closed and eyes-open EEG
  Variations in EEG brain connectivity, interhemispheric and frontoparietal connectivity (measured by band coherence, synchronicity likelihood, phase lag index), characteristic path and clustering coefficient (band coherence, synchronicity likelihood) in resting state (eyes-closed/open) in resting state eyes-closed/open EEG in DS compared to TD subjects.
Differences in cross-frequency coupling between DS and TD group | During resting state EEG, and while performing the auditory and the cognitive tasks
  Variations in cross-frequency coupling (theta-gamma coupling) during the resting state, the auditory and the cognitive tasks in DS compared to TD subjects.
Differences in Higuchi fractal dimension, small-world, characteristic path, and clustering coefficient between DS and TD group | During resting state eyes-closed and eyes-open EEG
  Variations in Higuchi fractal dimension, small-world, characteristic path, and clustering coefficient in DS compared to TD subjects.
Differences in plasma concentrations of endocannabinoids between DS and TD group | At baseline
  Variations in plasma concentrations of endocannabinoids (AEA and 2AG) in DS compared to TD subjects.
Differences in plasma concentrations of the neurosteroid pregnenolone between DS and TD group | At baseline
  Variations in plasma concentrations of the neurosteroid pregnenolone in DS compared to TD subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael de la Torre Fornell, PharmD, PhD, Principal Investigator — IMIM (Hospital del Mar Medical Research Institute)
Locations (1):
- IMIM (Hospital del Mar Medical Research Institute), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No